CLINICAL TRIAL: NCT05181267
Title: Effects of Intermittent Fasting on Insulin Resistance, Cardiac Metabolism, and Cerebral Perfusion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KETO-FAST
Record Dates: First submitted 2021-12-01; First posted 2022-01-06 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Insulin Resistance
Keywords: intermittent fasting; ketone bodies; obesity; cardiac substrate metabolism; insulin resistance; cerebral perfusion
MeSH Terms: conditions — Obesity; Insulin Resistance; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a randomized, controlled crossover study with 16 insulin-resistant subjects with overweight (BMI: 28-40 kg/m2) aged 55-70 years. Subjects must go through two study periods of each three weeks, where the interventions are alternate-day fasting (ADF) and Western diet (no restrictions), respectively, in random order. A washout period of one week follows the first study period before subjects cross over to the second study period. After each study period, subjects undergo a study day with PET scans and various laboratory examinations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent fasting (Experimental): Three weeks of alternate-day fasting.
  Interventions: Dietary Supplement: Intermittent fasting
- Western diet (No Intervention): Three weeks of normal Western diet (no restrictions).

INTERVENTIONS:
Dietary Supplement: Intermittent fasting — Subjects fast from after dinner and throughout the next day, i.e., 36 hours of fasting, after which they are allowed to eat as usual until dinner the same day. Then they fast again for 36 hours, and this regimen will continue for three entire weeks.
  Other Names: Alternate-day fasting
  Arms: Intermittent fasting

SUMMARY:
The overall purpose of the study is to investigate whether three weeks of intermittent fasting (alternate-day fasting, (ADF)) result in a more pronounced "metabolic shift" towards the use of ketone bodies than three weeks of Western diet. The investigators will use state-of-the-art PET/CT tracer techniques and well-established steady state kinetics methods for glucose and fatty acids. The study results will provide new insights into the physiological basis of the potential cardio-protective effects of ketone bodies during ADF and will determine whether ADF can help prevent and treat heart failure.

Ketone bodies are produced in the liver as an alternative fuel when blood glucose levels are low, as can be seen with various types of diets or after strenuous exercise. The energy produced by breaking down ketone bodies has been shown to require less oxygen than breaking down glucose and fatty acids. In a previous study, the investigators observed that ketone bodies act as a kind of "super fuel" for the heart and improve the heart's energy utilization. It is still unknown how high ketone levels are needed to see these cardio-protective effects. As patients with insulin resistance and/or heart failure have a lower glucose uptake in cardiac tissue, and as energy production by the breakdown of fatty acids is oxygen-demanding, an elevated level of blood ketones can therefore potentially reduce the morbidity seen in patients with type 2 diabetes and ischemic heart disease.

PET/CT is a non-invasive well-established imaging modality suitable for tracking the fate of metabolites, as most substances or metabolites can be labeled by a suitable PET isotope. PET has sufficient spatial and temporal resolution to enable direct quantification of e.g. uptake and oxidation rates and has been successfully used by the investigators' department to assess heart efficiency, oxygen consumption, and fatty acid metabolism. Currently, the investigators are in the process of validating the PET tracer 11C-beta-hydroxybutyrate (11C-3-OHB) as a radio tracer for human studies. The tracer will be able to detect changes in biodistribution and kinetics of ketone bodies during both Western diets and ADF.

The subjects must go through two study periods of each 3 weeks in which the intervention is western diet (no restrictions) and intermittent fasting (fasting every other day), respectively. After both study periods, there will be an examination day with PET scans and various laboratory examinations.

DETAILED DESCRIPTION:
Background

Ketone bodies are produced in the liver as an alternative fuel when blood glucose levels are low, such as during high-fat low-carb diets, prolonged calorie restriction, or after strenuous exercise. Ketone bodies from the blood are easily absorbed by energy-consuming tissues such as the heart and the brain, where they are oxidized to produce energy in the form of adenosine triphosphate (ATP).

ATP production by oxidation of ketone bodies requires less oxygen per mole of ATP produced than fatty acid oxidation, and therefore, ketone bodies have been called a "super fuel". As patients with insulin resistance and/or heart failure are characterized by a decreased glucose uptake into the heart tissue, and as ATP production by fatty acid oxidation is oxygen-demanding, an elevated level of ketone bodies in the blood (hyperketonemia) therefore has the potential to reduce myocardial ischemia-related morbidity in individuals with insulin resistance, type 2 diabetes, and ischemic heart disease.

The investigators have previously demonstrated that the heart easily switches from glucose to ketone body consumption when ketone body levels are rapidly increased by an infusion, resulting in a 50% reduction in cardiac glucose consumption. In addition to the presumed beneficial effects on oxygen consumption, the investigators also observed a marked increase in cardiac output; findings which they subsequently confirmed with studies of heart failure patients in which a linear dose-response relationship between the level of ketone bodies and cardiac output was observed.

Calorie restriction (CR) is a term used for continuous energy restriction representing 30% or more of the basic energy requirement. CR has consistently and not surprisingly been shown to promote weight loss but also reduce the risk of cardiovascular disease. However, CR is associated with several side effects, including decreased bone mass and bone mineral density, and relative leukopenia, which can potentially increase the risk of infections. In addition, individuals undergoing CR diets complain of hunger, irritability, and decreased concentration. This results in a low, and often non-lasting, long-term success rate.

Intermittent fasting (IF) is a term that describes different dietary patterns that involve complete or partial limitation of energy intake at different time periods and at specific time intervals. IF has been shown to result in roughly the same beneficial effects as CR. IF causes a weight loss, as the calorie intake on the days without fasting does not fully compensate for the calorie deficit on days with fasting. Various forms of IF exist, including 5:2 diet, complete alternate-day fasting (ADF), modified ADF, and time-restricted feeding. However, it is only during the 5:2 diet and the complete ADF that the fasting periods exceed 20 hours, which has major consequences for the hormonal and metabolic environment of the fasting persons. Fasting for 20 hours or more results in low blood glucose levels and an almost complete inhibition of insulin secretion. It stimulates ketogenesis in the liver and lipolysis in adipose tissue with the release of fatty acids as a substrate for the formation of ketones. This is the so-called "metabolic shift" that most individuals in the Western world, including people on the CR diet, rarely experience. The metabolic shift during IF has been shown to improve insulin sensitivity and to provide weight loss; even to a greater extent than during CR. Overall, it seems that the same benefits of CR can be achieved by exercising an IF regimen, but only the latter triggers hyperketonemia with the associated, presumed, cardiac benefits. An increased level of ketone bodies has also been shown to improve cognitive function in patients with impaired cognition or mild Alzheimer's disease. This can potentially be explained by an increased perfusion in the blood vessels of the brain, which is seen in ketosis.

PET/CT is a non-invasive imaging modality that is well-established in oncological staging and treatment monitoring. The technique is also suitable for tracking the fate of metabolites, as most substances or metabolites can be labeled by a suitable PET isotope. PET has sufficient spatial and temporal resolution to enable direct quantification of e.g., uptake and oxidation rates and has been successfully used by the investigators' department to assess heart efficiency, oxygen consumption, and fatty acid metabolism. Currently, the investigators are in the process of validating the newly developed ketone PET tracer 11C-3-OHB as a radiotracer for human studies. The tracer will make it possible to detect changes in biodistribution and kinetics of ketone bodies during both Western diets and during fasting regimens such as ADF.

Purpose

The aim of the study project is to investigate whether intermittent fasting in the form of three weeks of ADF improves insulin resistance, as well as cardiac pump function and substrate metabolism compared to three weeks of regular Western diet. In addition, the investigators wish to examine the perfusion in the brain, which has been shown to be increased during ketosis. State-of-the-science PET/CT tracer techniques and well-established steady-state kinetics methods for glucose and fatty acids will be applied. The study results will help clarify whether ADF should be recommended in the non-pharmacological prophylaxis and treatment of insulin resistance, type 2 diabetes, and heart failure, as well as a possible increase in brain perfusion improving the cognitive function in these patients.

Specific aims:

1. To measure cardiac uptake and metabolism of hydroxybutyrate after ADF versus Western diet (11C-3-OHB PET)
2. To measure myocardial perfusion and flow reserve after ADF compared to Western diet (15O-dihydrogen monoxide (H2O) PET)
3. To determine the effect of ADF compared to Western diet on insulin sensitivity in skeletal muscle, liver, and adipose tissue (hyperinsulinemic-euglycemic clamp)
4. To measure myocardial external efficiency (MEE) after ADF compared to Western diet (11C-acetate PET)
5. To measure cardiac metabolism of fatty acids and glucose after ADF compared to Western diet (11C-palmitate and fluorine-18-fluorodeoxyglucose (18F-FDG) PET, respectively)
6. To measure cerebral perfusion after ADF versus Western diet (15O-H2O PET)
7. To assess insulin signaling in skeletal muscle and adipose tissue after ADF compared to Western diet (muscle and fat biopsies)
8. To characterize daily time-related changes in fatty acids, glucose, and ketone bodies during three weeks of ADF

Methods

The study will be conducted as a randomized, controlled crossover study with 16 insulin-resistant subjects with overweight (BMI: 28-40 kg/m2) aged 55-70 years.

Before initiating the study, the subjects will go through a screening visit in undisturbed surroundings at Aarhus University Hospital, where the subjects can give their informed consent if they wish to participate in the study. Beforehand, they are informed that they have the right to bring an attendant to the visit. After signed consent, there will be a conversation about the subjects' health, blood samples will be taken, height, weight and blood pressure measured, and an ECG performed. In addition, a transthoracic echocardiography will be performed to rule out structural heart disease.

If the inclusion criteria are still met and the exclusion criteria are not, subjects will be instructed to fast for 36 hours from 7 p.m. on day -3 as a run-in period to make sure they can meet the time schedule for fasting. After this, they must go through two study periods of each three weeks, where the interventions are ADF and Western diet (no restrictions), respectively, in random order. A washout period of one week follows the first study period before subjects cross over to the second study period. The subjects will approx. once a week be contacted by telephone to ensure compliance to the ADF regimen.

At the start of the first study period and at the end of each study period, blood samples will be taken, and a 24-hour urine sample will be performed, where all urine produced in one day will be collected by the subject in a plastic can for the purpose. The urine is destroyed after the analysis. Subjects will also be asked about risk factors for osteoporosis.

In both study periods, the concentration of ketone bodies will be measured by the subjects twice daily (7 a.m. and 7 p.m.) with ketone strips on a hand-held glucose meter at home. If subjects increase less than 0.3 millimolar (mM) in ketone body levels after one week of ADF (as an expression of non-compliance with the diet), they will drop out of the study without further follow-up. At the end of each study period, the subjects will have a ketone profile made with 6 measurements/day over three days.

After each study period, subjects undergo an examination day with PET/CT scans and various laboratory examinations. For 72 hours up to the examination days, subjects will be asked to avoid alcohol and strenuous physical activity. They will have their physical activity monitored with an activity meter (FitBit Charge 2), as well as blood pressure/vascular stiffness with a 24-hour blood pressure monitor. In addition, they will be asked to fast from 10 p.m. the evening before both examination days.

ELIGIBILITY:
Inclusion Criteria:

* Age: 55-70 years
* BMI: 28-40 kg/m2

Exclusion Criteria:

* Any drug that, in the investigator's opinion, may affect the study
* HbA1c > 48 mmol/mol
* Known heart failure, previous blood clots, or other heart disease that, in the investigator's opinion, may affect the study, including abnormal ECG and/or echocardiography with evidence of structural heart disease
* Liver disease (ALAT > 3 x of upper normal range), renal failure (eGFR < 60 ml/min), anaemia (Hb < 6.5), current or previous malignant disease which, in the investigator's opinion, may affect the study
* Current alcohol abuse (> 21 items per week)
* Blood donation within the last 3 months before the study day
* Participation in studies/examinations involving radioactive isotopes within the last 6 months
* Claustrophobia

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac uptake and metabolism of hydroxybutyrate | The PET/CT scan will be performed on the study day after each 3-week study period (day 22 and 51).
  Change in cardiac uptake and metabolism of hydroxybutyrate after ADF versus Western diet will be measured with 11C-3-OHB PET/CT.
Change in myocardial perfusion and flow reserve | The PET/CT scan will be performed on the study day after each 3-week study period (day 22 and 51).
  Change in myocardial perfusion and flow reserve after ADF compared to Western diet will be measured with 15O-H2O PET/CT.
Change in insulin sensitivity in skeletal muscle, liver and adipose tissue | The clamp will be performed on the study day after each 3-week study period (day 22 and 51).
  Effect of ADF compared to Western diet on insulin sensitivity in skeletal muscle, liver, and adipose tissue will be measured by a hyperinsulinemic-euglycemic clamp. Subjects will undergo the clamp during the study day. The amount of infused glucose during the clamp will act as a measure of the subjects' insulin sensitivity/resistance.
Change in cardiac uptake and metabolism of fatty acids | The PET/CT scan will be performed on the study day after each 3-week study period (day 22 and 51).
  Change in cardiac uptake and metabolism of fatty acids after ADF compared to Western diet measured with 11C-palmitate PET/CT.
Change in cardiac uptake and metabolism of glucose | The PET/CT scan will be performed on the study day after each 3-week study period (day 22 and 51).
  Change in cardiac uptake and metabolism of glucose after ADF compared to Western diet measured with 18F-FDG PET/CT.
Change in cerebral perfusion | The PET/CT scan will be performed on the study day after each 3-week study period (day 22 and 51).
  Change in cerebral perfusion after ADF versus Western diet measured with 15O-H2O PET/CT.

SECONDARY OUTCOMES:
Changes in insulin signaling in skeletal muscle and adipose tissue | The biopsies will be performed on the study day after each 3-week study period (day 22 and 51).
  Proteins involved in insulin signaling and lipolysis will be determined by Western blot analysis of muscle and adipose tissue biopsies.
Changes in circulating concentrations of free fatty acids, cholesterol, glucose, and hemoglobin | Blood samples will be taken at the screening visit (before day -3) and on the study day after each 3-week study period (day 22 and 51).
  Measured in blood samples [mmol/L]
Changes in circulating concentrations of lactate dehydrogenase, glucagon, hydroxybutyrate, gastric inhibitory peptide, and glucagon-like peptide-1, alanine transaminase, alkaline phosphatase, and erythropoietin. | Blood samples will be taken at the screening visit (before day -3) and on the study day after each 3-week study period (day 22 and 51).
  Measured in blood samples [units/L]
Changes in circulating concentrations of C-reactive protein. | Blood samples will be taken at the screening visit (before day -3) and on the study day after each 3-week study period (day 22 and 51).
  Measured in blood samples [mg/L]
Change in myocardial external efficiency (MEE) | The PET/CT scan will be performed on the study day after each 3-week study period (day 22 and 51).
  Change in myocardial external efficiency (MEE) after ADF compared to Western diet will be measured with 11C-acetate PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Mette LG Kjærulff, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark